CLINICAL TRIAL: NCT02344173
Title: ABLATOR Ablation Observational Registry
Acronym: ABLATOR
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD_723
Record Dates: First submitted 2015-01-13; First posted 2015-01-22 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this registry is to assess the performance and clinical effectiveness of a combination of SJM mapping and ablation products in the treatment of subjects with atrial fibrillation (AF).

DETAILED DESCRIPTION:
The objectives of this registry are the following:

* To confirm patient safety as part of the post market surveillance study.
* To assess performance of a combination of SJM products during procedures.
* To assess the learning curve with a combination of SJM products.
* To collect operator feedback on a combination of SJM products.

All patients from participating sites who are indicated for an atrial fibrillation ablation procedure and willing to provide written Informed Consent may be enrolled in this registry.

In order to ensure a minimum level of uniformity across site practices and to enable comparison of acute and long-term effectiveness as well as procedure efficiency according to technique used, a combination of 2 types of devices from the pre-specified list must be used to be eligible in this registry.

ELIGIBILITY:
Inclusion Criteria:

All patients who are indicated for an atrial fibrillation ablation procedure.

Exclusion Criteria:

Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are indicated for an atrial fibrillation ablation procedure.
Sampling Method: Non-Probability Sample
Enrollment: 2035 (Actual)
Dates: Start 2014-11; Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- Allgemeines Krankenhaus Linz, Linz, Austria
- Belgium (3):
  - AZ Middelheim, Antwerp
  - Jessa Ziekenhuis, Hasselt
  - CHR Citadelle, Liège
- Canada (4):
  - Foothills Medical Center, Calgary
  - QE II Health Sciences, Hailfax
  - Royal Jubilee hospital, Newmarket
  - Institut de Cardiologie de Quebec (Hôpital Laval), Québec
- China (6):
  - Fuwai Heart Hospital & Cardiovascular Institute, Beijing
  - Third Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Chengdu
  - Sir Run Run Shaw Hospital, Hangzhou
  - Prince of Wales Hospital, Hong Kong
  - Ningbo 1st. Hospital, Ningbo
- FN U sv. Anny v Brno, Brno, Czechia
- France (5):
  - Clinique Rhône-Durance-Avignon, Avignon
  - CHU Brest, Brest
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHRU Lille, Lille
  - Clinique Pasteur, Toulouse
- Germany (12):
  - Zentralklinikum Bad Berka, Bad Berka
  - Herz- und Gefässzentrum Bad Bevensen, Bad Bevensen
  - Kerckhoff Klinik, Bad Nauheim
  - Vivantes Klinikum Am Urban, Berlin
  - Immanuel Klinikum Bernau - Herzzentrum Brandenburg, Bernau
  - Universitätsklinikum Köln, Cologne
  - Herz- und Gefässzentrum am Krankenhaus Neu-Bethlehem, Göttingen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Herzzentrum Leipzig, Leipzig
  - Klinikum Ludwigshafen, Ludwigshafen
  - Märkische Kliniken GmbH Klinikum Lüdenscheid, Lüdenscheid
  - Kliniken Maria Hilf, Mönchengladbach
- India (4):
  - Fortis Hospital Limited, Bangalore
  - Medanta - The Medicity Hospital, Gūrgaon
  - Escorts Heart Institute and Research Centre, New Delhi
  - Christian Medical College & Hospital, Vellore
- Italy (6):
  - Ospedale Cardinal Massaia, Asti, Piedmon
  - Ospedale San Giovanni di Dio - Torregalli, Florence, Tuscany
  - Ospedale SS Antonio e Biagio, Alessandria
  - Fondazione Giovanni Paolo II, Campobasso
  - Ospedale Spirito Santo, Pescara
  - Ospedale San Filippo Neri, Roma
- Netherlands (3):
  - Catharina Hospital, Eindhoven
  - Erasmus Rotterdam, Rotterdam
  - Haga Hospital, The Hague
- Portugal (3):
  - Hospital Santa Cruz, Carnaxide
  - Hospital Santa Maria, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Prince Sultan Cardiac Center, Riyadh, Saudi Arabia
- South Korea (4):
  - Yeungnam University Medical Center, Daegu
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Health System, Seoul
- Spain (5):
  - Hospital general Universitario de Alicante, Alicante
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital do Meixoeiro, Vigo
- United Kingdom (4):
  - Royal Bournemouth Hospital, Bournemouth
  - Royal Sussex County Hospital, Brighton
  - Castle Hill Hospital, Hull
  - Leeds General Infirmary, Leeds

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Subjects: Subjects enrolled in the registry were already planned to undergo an ablation procedure for AF (including both first ablation and repeat ablations). Subjects were considered enrolled upon providing written informed consent.
Period: Enrollment
Arm/Group | All Enrolled Subjects
Started | 2035
Completed | 2035
Not Completed | 0
Period: Procedure
Arm/Group | All Enrolled Subjects
Started | 2035
Completed (Ablation procedure performed.) | 2028
Not Completed | 7
Not completed — Ablation Procedure Not Performed | 7
Period: 12-month Visit
Arm/Group | All Enrolled Subjects
Started | 2028
Completed | 1932
Not Completed | 96
Not completed — Death | 8
Not completed — Withdrawal by Subject | 30
Not completed — Lost to Follow-up | 58

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 2035
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data for 1 patient is missing.
  years
    number analyzed (Participants) | 2034
    (all) | 61.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data is missing for 3 patients.
  Participants
    number analyzed (Participants) | 2032
    Female | 639
    Male | 1393
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Indication for procedure [Count of Participants; unit: Participants] — Population: Data is missing for 7 patients.
  Participants
    number analyzed (Participants) | 2028
    Paroxysmal AF | 1151
    Persistent AF | 746
    Permanent AF | 131
Had Prior AF Ablation [Count of Participants; unit: Participants] — Population: Data missing for 7 patients.
  Participants
    number analyzed (Participants) | 2028
    Yes | 1581
    No | 447
Percentage of Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: %] — Population: Measure Analysis Population Description: Data not collected from all patients.
  %
    number analyzed (Participants) | 1178
    (all) | 58.7 (9.4)
Left Atrial Diameter [Mean (Standard Deviation); unit: mm] — Population: Data not collected from all patients.
  mm
    number analyzed (Participants) | 1251
    (all) | 42.5 (11.2)
Left Atrial Volume [Mean (Standard Deviation); unit: mL] — Population: Data not collected from all patients.
  mL
    number analyzed (Participants) | 476
    (all) | 76 (39.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Achieved Freedom From AF/AFL/AT (Atrial Fibrillation/Atrial Flutter/Atrial Tachycardia) With or Without the Use of Anti-arrhythmic Drugs After a 3-month Blanking Period.
Description: Freedom from AF/AFL/AT (atrial fibrillation/atrial flutter/atrial tachycardia) with or without the use of anti-arrhythmic drugs after a 3-month blanking period. Repeat ablations during the 3-month blanking period do not count as effectiveness failures. A repeat ablation procedure after the 3-month blanking period is counted as an effectiveness failure.
Time Frame: 12 months post procedure
Population: Subjects that completed 12-month visit
Measure: Count of Participants; unit: Participants
Groups:
- Per-Protocol: Patients that were enrolled, received RF ablation therapy, and completed 12-month follow-up
Arm/Group | Per-Protocol
Number analyzed (Participants) | 1932
Participants | 1297

2. Primary Outcome: Number of Subjects That Achieved Freedom From AF/AFL/AT (Atrial Fibrillation/Atrial Flutter/Atrial Tachycardia) With or Without the Use of Anti-arrhythmic Drugs After a 3-month Blanking Period.
Description: as for outcome 1
Time Frame: 12 months post procedure
Population: Treated Subjects
Measure: Count of Participants; unit: Participants
Groups:
- Treated Subjects: Patients that were enrolled and received RF ablation therapy.
Arm/Group | Treated Subjects
Number analyzed (Participants) | 2028
Participants | 1297

3. Primary Outcome: Number of Subjects That Experienced 1 or More Procedure and/or Device-related Cardiovascular SAE/SADEs.
Description: Procedure and/or Device-Related Cardiovascular SAE/SADEs. This registry collected information about adverse events deemed of cardiovascular origin ("Cardiovascular Serious Adverse Event") with the potential of leading to:
  * Death
  * A serious deterioration in the health of the subject
  * Fetal distress, fetal death or a congenital abnormality or birth defect
  A planned hospitalization for a pre-existing condition was not considered a serious adverse event. Reporting of non-serious events and non-cardiovascular events was not required.
Time Frame: 12 months post procedure
Population: Enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 2035
Participants | 43

ADVERSE EVENTS:
Time Frame: SAE/SADE information was collected from the time of enrollment through 12 months (+/- 30 day visit window)
Description: Only SAEs deemed to be of a cardiovascular origin were reportable in ABLATOR. A planned hospitalization for a pre-existing condition was not considered an SAE. Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 8/2035
Serious Adverse Events (participants affected / at risk) | 356/2035
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=2035)
Abnormal ECG (Cardiac disorders) | 5 (5)
Angina (Chest Pain) (Cardiac disorders) | 11 (11)
Arrhythmia (Cardiac disorders) | 249 (304)
Atrio-esophageal fistula (Gastrointestinal disorders) | 1 (1)
AV Fistula (Vascular disorders) | 1 (1)
Complete Heart Block (Cardiac disorders) | 3 (3)
Death (General disorders) | 2 (2)
Exacerbation of Pre-Existing Atrial Fibrillation (Cardiac disorders) | 21 (26)
Heart Block (Cardiac disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 5 (5)
Hypotension (Vascular disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 2 (2)
Obstruction/Perforation/Damage of The Vascular System (Vascular disorders) | 2 (2)
Other (General disorders) | 31 (36)
Palpitation (Cardiac disorders) | 7 (7)
Pericardial Effusion Without Tamponade (Cardiac disorders) | 6 (7)
Pericardial Effusion/Cardiac Tamponade (Cardiac disorders) | 14 (14)
Pericarditis (Cardiac disorders) | 4 (4)
Pulmonary Edema (Cardiac disorders) | 1 (1)
Pulmonary Vein Stenosis (Vascular disorders) | 1 (1)
Pulmonary Vein Thrombus (Vascular disorders) | 1 (1)
Sinus Node Dysfunction (Cardiac disorders) | 8 (8)
Stroke/cerebral vascular accidents (Nervous system disorders) | 5 (5)
Vascular Access/Bleeding Complications (Vascular disorders) | 9 (10)
Ventricular Arrhythmia Requiring Defibrillation (Cardiac disorders) | 2 (2)
Vessel Wall/Valvular Damage or Insufficiency (Vascular disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
SAEs were adjudicated by the sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT02344173/Prot_SAP_000.pdf